CLINICAL TRIAL: NCT00003810
Title: A Phase II Study of Gemcitabine and Docetaxel in Pancreatic Adenocarcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Locally Advanced or Metastatic Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066955; ECOG-1298
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Docetaxel; Gemcitabine

INTERVENTIONS:
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more that one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine and docetaxel in treating patients who have locally advanced or metastatic cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate of patients with pancreatic adenocarcinoma treated with combination gemcitabine and docetaxel. II. Determine the toxicity profile of this combination therapy in these patients. III. Assess the survival rate of these patients.

OUTLINE: Patients receive docetaxel IV over 1 hour followed by gemcitabine IV over 30 minutes. Patients receive treatment every other week for 8 weeks (4 courses). Patients may continue treatment in the absence of unacceptable toxicity or disease progression. Patients are followed every 12 weeks until death.

PROJECTED ACCRUAL: This study will accrue approximately 10 patients per month for a maximum of 33 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma or poorly differentiated carcinoma of the pancreas Metastatic disease with at least 1 bidimensionally measurable lesion OR Locally advanced disease that is either recurrent or not amenable to surgery Measurable disease outside of prior radiation port or disease progression within the port

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1500/mm3 Platelet count at least 125,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) SGOT no greater than 2.5 times ULN (less than 3 times ULN if liver metastases) Renal: Creatinine no greater than ULN Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic disease At least 1 year since prior adjuvant chemotherapy Prior chemoradiotherapy as initial therapy allowed Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics See Chemotherapy At least 4 weeks since prior radiotherapy Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08-11 (Actual); Primary Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Shepard, MD, Study Chair — University of Virginia
Locations (10):
- United States (10):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Shepard RC, Levy DE, Berlin JD, Stuart K, Harris JE, Aviles V, Thomas JP, Benson AB 3rd. Phase II study of gemcitabine in combination with docetaxel in patients with advanced pancreatic carcinoma (E1298). A trial of the eastern cooperative oncology group. Oncology. 2004;66(4):303-9. doi: 10.1159/000078331. PMID 15218298
- [Result] Ryan DP, Kulke MH, Fuchs CS, Grossbard ML, Grossman SR, Morgan JA, Earle CC, Shivdasani R, Kim H, Mayer RJ, Clark JW. A Phase II study of gemcitabine and docetaxel in patients with metastatic pancreatic carcinoma. Cancer. 2002 Jan 1;94(1):97-103. doi: 10.1002/cncr.10202. PMID 11815964
- [Result] Shepard RC, Levy D, Stuart K, et al.: Pancreatic cancer: biweekly gemcitabine/docetaxel chemotherapy. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-614, 2001.